CLINICAL TRIAL: NCT05618379
Title: Adult Patients With Spinal Muscular Atrophy in China: A Nationwide Registry
Brief Title: Adult Spinal Muscular Atrophy (SMA) China Registry
Status: Active, not recruiting | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: CN-SMG-11772
Record Dates: First submitted 2022-10-20; First posted 2022-11-16 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Muscular Atrophy, Spinal
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DMT Treated Participants: Participants with SMA who received prior treatment with DMTs including nusinersen will be followed prospectively for up to 60 months and the available data is collected retrospectively.
- Untreated Participants: Participants with SMA who received no treatment will be followed prospectively for up to 60 months.

SUMMARY:
The primary objective of the study is to describe the natural history and utilization of disease modifying therapy (DMT) among adult Chinese participants with SMA linked to chromosome 5q (5q-SMA).

ELIGIBILITY:
Key Inclusion Criteria:

-Genetically confirmed 5q-SMA.

Key Exclusion Criteria:

-Other types of SMA (non 5q-SMA).

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult participants with 5q-SMA will be enrolled to obtain information on both the natural history of the disease and effectiveness and safety of DMTs.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-01-06 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Characterized by Natural History of 5q-SMA Observed Among Adult Chinese Participants | Up to 60 Months
  The natural history characteristics will include the categories of the evolution of the patient's condition over the time of data collection from the registry, to describe the natural history of the disease in a real-life situation.
Number of Participants Characterized by Utilization of Disease Modifying Therapies (DMTs) of 5q-SMA Observed Among Adult Chinese Participants | Up to 60 Months
  The DMT utilization characteristics will include the categories of the evolution of the DMT treated patient's condition over the time of data collection from the registry, to describe the utilization of DMTs of adult SMA patients in a real-life situation.

OTHER OUTCOMES:
Time to Mortality | Up to 60 Months
  Time interval between baseline and death.
Number of Participants With Clinical Characteristics | Up to 60 Months
  Clinical characteristics will include categories of motor function, motor measures, pulmonary function, clinical observations, nutrition, electrophysiology, biomarkers and categories of patient reported measures
Number of Participants with Hospitalization | Up to 60 Months
Number of Participants With Comorbidities | Up to 60 Months
Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAEs) | Up to 60 Months
  An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. SAE is any untoward medical occurrence that at any dose results in death, in the view of the investigator, places the participant at immediate risk of death (a life-threatening event), requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in a congenital anomaly/birth defect or is a medically important event.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (12):
- China (12):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - The First People's Hospital of Yunnan Province, Kunming, Yun'nan

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

REFERENCES:
- [Derived] Dai Y, Yao X, Zhu W, Zhao Y, Shang H, Chen J, Meng Q, Liu Y, Chen W, Yu L, Shen L, Hong D, Chen K, Zhang L, Mai M, Cui L. Effectiveness and Safety of Nusinersen Among Adults with 5q-Spinal Muscular Atrophy: A Multicenter Disease Registry in China. Adv Ther. 2025 Dec 29. doi: 10.1007/s12325-025-03475-2. Online ahead of print. PMID 41461996